CLINICAL TRIAL: NCT02257944
Title: Assessing and Reducing Risk of Violent Re-Injury Among Victims of Urban Violence: A Randomized Clinical Trial
Brief Title: Assessing and Reducing Risk of Violent Re-Injury Among Victims of Urban Violence
Acronym: VOV-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Conrad, Erich J., M.D. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSUHSC-8692
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Violence
MeSH Terms: interventions — Motivational Interviewing; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing (Experimental): Receive brief hospital-based intervention
  Interventions: Behavioral: Motivational Interviewing
- Treatment as Usual (Other): Treatment as Usual
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Motivational Interviewing — Brief hospital-based intervention, rooted in motivational interviewing
  Arms: Motivational Interviewing
Other: Treatment as Usual — treatment as usual
  Arms: Treatment as Usual

SUMMARY:
The purpose of the study is to develop a program to help people to lower their chances of being violently injured again.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-65 years
* intentionally injured in community violence.
* admitted to a Level 1 trauma center
* able to provide voluntary informed consent

Exclusion Criteria:

* under the age of 18 or over the age of 55.
* not fluent in the English language
* patients with suspected mental retardation or active psychosis as determined by brief clinical screen.
* patients currently in legal detention status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Risk Factors for Violence | 3 months
  interview of risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Erich J Conrad, MD, Principal Investigator — LSUHSC Trauma Psychiatry Reserach Unit